CLINICAL TRIAL: NCT05989685
Title: Psychometric Validation of the Camouflaging Autistic Traits Questionnaire (CAT-Q/DE) in a German Population of Autistic and Non-autistic Adolescents.
Brief Title: Psychometric Validation of the Camouflaging Autistic Traits Questionnaire
Acronym: CAT-Q/DE
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Johannes Boettcher, Dr., Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: LPEK-0659
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Camouflaging; Late diagnosis; Adolescents
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Adolescents between the ages of 13-21 who meet diagnostic criteria for an autism spectrum disorder.
- Control group: Adolescents aged 13-21 years without a lifetime psychiatric diagnosis.

SUMMARY:
For many affected individuals, despite impairment and distress, autism spectrum disorder (ASD) is recognized and diagnosed late, in school age, adolescence, or even in adulthood, which could be due, among other things, to the use of compensatory strategies such as so-called "camouflaging" by the respective individual. In order to better investigate and quantify these adaptive and compensatory strategies of individuals with autism, the Camouflaging Autistic Traits Questionnaire (CAT-Q) has recently been developed and validated in the English-speaking world. The CAT-Q is designed to assess the extent of camouflaging behavior, in which autistic individuals consciously or unconsciously attempt to conceal or attenuate their autistic traits in order to better adapt to social situations. So far, however, there is no German-language questionnaire that can be used to validly assess camouflaging. The aim of the planned research project is to psychometrically validate the CAT-Q in German-speaking adolescents aged 13-21 years. The validation of the CAT-Q represents an important basis for further research on the construct camouflaging and can subsequently contribute to an improvement of diagnostics as well as support the development of individual treatment approaches.

ELIGIBILITY:
Inclusion Criteria study group:

- patients who meet the principal diagnosis of ASD, which includes atypical autism (ICD-10: F84.1) and Asperger syndrome (ICD-10: F84.5), and are between the ages of 13 and 21 years old.

Exclusion Criteria study group:

* Dementia / below average cognitive abilities (IQ < 85)
* lack of German language skills
* severe visual or hearing impairment (uncorrected)

Inclusion Criteria control group:

- Adolescents who do not have a lifetime principal diagnosis of a psychiatric disorder (ICD-10-GM-2016: F10 - F69) and are between 13 and 21 years old.

Exclusion Criteria Control Group:

* dementia / below average general cognitive ability (IQ < 85)
* lack of German language skills
* severe impairment of vision or hearing (not corrected).

Ages: 13 Years to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients treated at the Department of Child and Adolescent Psychiatry, Psychotherapy, and Psychosomatics at the UKE and the joint practice - KJP Praxis Hoheluft, as well as other participants who meet the diagnostic criteria of an autism spectrum disorder will be included in the study. Interrater reliability between the sites will be recorded and assessed to ensure that the diagnostic criteria of an autism spectrum disorder are applied consistently between the two sites. The control group will be recruited through Bilendi-Respondi, a market research service provider.
Sampling Method: Probability Sample
Enrollment: 622 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Camouflaging | 3-4 minutes
  Camouflaging Autistic Traits Questionnaire (CAT-Q; Hull et al., 2019) is a quantitative measure of camouflaging. The CAT-Q can be used as a self-report and parent report version. The CAT-Q was constructed to be appropriate for both autistic and non-autistic populations (Hull et al., 2019). The instrument includes 25 items that are answered on a seven-point Likert scale.

SECONDARY OUTCOMES:
Autistic Traits | 3 minutes
  The Social Responsiveness Scale (SRS-16; Constantino et al., 2003) is a quantitative measure of autistic traits in children, adolescents, and adults. The SRS-16 (Sturm et al., 2017) is a 16-item parent questionnaire assessing social, communicative, and rigid behaviors in children and adolescents in terms of a dimensional diagnosis of autism.
Mental health | 4 minutes
  The Strengths and Difficulties Questionnaire (SDQ; Goodman, 1997) is one of the most frequently used methods for assessing mental health in children and adolescents from a self- and parent perspective. In addition to the version for children and adolescents, there is also a version for adults, the SDQ 18+. The SDQ assesses mental health problems and resources of children and adolescents with 5 items each on five subscales: behavioral problems, emotional problems, hyperactivity, peer problems, and prosocial behavior. It has good psychometric properties, is economical, and has been widely used in research (Goodman, 2001).
Symptoms of depression | 1 minutes
  The Patient Health Questionnaire scale 9 (PHQ-9; (Kroenke et al., 2001), is a self-report questionnaire designed to assess the severity of depressive disorder in adolescents and adults. The PHQ-9 has been shown to display good psychometric properties and has been validated in autistic adolescents and adults (Arnold et al., 2020).
Symptoms of anxiety | 1 minutes
  The Generalized Anxiety Disorder scale 7 (GAD-7; Spitzer et al., 2006), is a self-report questionnaire designed to assess the severity of anxiety in adolescents and adults. The GAD-7 has been validated in adolescent and adult populations, displaying good psychometric properties (Löwe et al., 2008). The GAD-7 is strongly correlated with anxiety measures including the Beck Anxiety Inventory (Spitzer et al., 2006) and provides a valid measure also of other anxiety disorders, e.g. social anxiety and panic disorder (Kroenke et al., 2007).
Stress | 1 minutes
  The Perceived Stress Scale (PSS-10; Schneider et al., 2020) is a 10-item questionnaire commonly used to assess stress levels in adolescents and adults 12 years and older. It assesses the extent to which a person has perceived life as unpredictable, uncontrollable, and overwhelming in the past month.
Loneliness | 1 minute
  3-item Loneliness Scale (Klein et al., 2021): Loneliness is also measured by the 3-item Loneliness Scale. The scale is an economic measure derived from the R-UCLA Loneliness Scale (Russell et al., 1980) that captures basic aspects of loneliness: A sense of isolation, disconnectedness, and not belonging. Items are rated on 5-point Likert scales. Responses are summed for a total score ranging from 0 to 12, with higher scores indicating higher levels of loneliness. Autism related adaptations of the instrument was made according to recent research (Grace et al., 2023).
Mentalizing | 1 minute
  The Reflective Function Questionnaire for Youth-5 (RFQ-Y; Sharp et al., 2022) measures mentalizing ability in adolescents. The English version showed satisfactory psychometric properties (Sharp et al., 2022).
Theory of Mind | 3-4 minutes
  The Frith-Happé Animations Test (Livingston et al., 2021), which represents interactions between triangles in animations, is an online instrument for measuring Theory of Mind (ToM). The web-based version of this test provides a quick and objective measurement of the construct ToM using multiple-choice questions. The instrument demonstrated good psychometric properties in a clinical as well as a non-clinical sample (Livingston et al., 2021).
Emotion Regulation | 1 minute
  The Difficulties in Emotion Regulation Scale (DERS; Gratz and Roemer, 2004) was used to measure difficulties in emotion regulation. Although there are different versions, this study we will use the short version with 8 items as suggested by Penner & Sharp, 2022. The DERS-8 has shown good psychometric properties (Penner & Sharp, 2022).
Parent-Adolescent Communication | 2-3 minutes
  The quality of dyadic Parent-Adolescent Communication was assessed with the German translation of the Parent-Adolescent Communication Scale (PACS; Barnes & Olson, 1982). The original measure consists of an adolescent and a parent version with 20 identical items that are rated on a scale from 1 ("strongly disagree") to 5 ("strongly agree"). The German version of the instrument has shown acceptable psychometric properties (Zapf & Boettcher, 2024)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Boettcher, Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Sarah Hohmann, Prof. Dr., Study Chair — Universitätsklinikum Hamburg-Eppendorf; Carola Bindt, Dr., Study Chair — Universitätsklinikum Hamburg-Eppendorf; Benno Schimmelmann, Prof. Dr., Study Chair — Universitäre Psychiatrische Dienste Bern
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- Available data/document: Statistical Analysis Plan — https://osf.io/dmyuq/files/osfstorage/67cb0a2098ee14b2b7fd7157 — Statistical Analysis Plan available in OSF.